CLINICAL TRIAL: NCT07075731
Title: Cervical and Endometrial Cancer Screening in Patients Seeking Gender-Affirming Hysterectomy
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2023LS213
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cancer Screening; Transgender; Gender Diverse Populations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard of Care Cancer Screening
  Interventions: Other: No intervention
- FDA approved self swab
  Interventions: Other: No intervention
- Mock self swab
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
This study aims to quantify the rates of cervical cancer screening and endometrial sampling prior to gender-affirming hysterectomy, assess the need for these tests in TGD individuals, and explore patient-centered options for these tests. By assessing the status of testing and correlation with hysterectomy pathology, this study will provide preliminary data on the current state of guideline-concordant care and provide initial evidence for the development of evidence-based guidelines in the future

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to provide voluntary written consent prior to the performance of any research related activity. Patients who can provide informed consent
* Able to understand, speak, read, and write in English
* Patients who have undergone hysterectomy, or plan to have a hysterectomy
* Patients who are transgender and gender diverse"

Exclusion Criteria:

* Opted out of research
* <18 years old
* Lacks capacity to consent/has diminished capacity to consent
* Cannot provide informed consent
* Those on the study's community advisory board

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone hysterectomy, or plan to have a hysterectomy. Patients who are transgender and gender diverse
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of cervical cancer screening and endometrial sampling in TGD individuals | Month 36
  Describe the rates of cervical cancer screening and endometrial sampling in TGD individuals undergoing hysterectomy in the MHealth Fairview System between January 2014-June 2024.
Whether HPV self-testing affects the rates of cervical cancer screening in TGD individuals | Month 36
  Describe the rates of cervical and endometrial cancer and their precursor lesions on pathology after hysterectomy that was undiagnosed prior to hysterectomy in TGD individuals in the MHealth Fairview System between January 2014-June 2024.

SECONDARY OUTCOMES:
how introducing the option of HPV self-testing affects the rates of cervical cancer screening in TGD individuals undergoing hysterectomy. | Month 36
  Assess how introducing the option of HPV self-testing affects the rates of cervical cancer screening in TGD individuals undergoing hysterectomy. Patients planning hysterectomy who are not up to date on cervical cancer screening will be offered standard cervical cancer screening or HPV self-testing. These participants will also be recruited to complete surveys and interviews. Patients who are up to date on cervical cancer screening prior to their hysterectomy consult will have the option to complete a mock self-swab or no testing. Participants who are up to date on cervical cancer screening will be surveyed regarding their experiences with cervical cancer screening and how the self-testing option impacts cervical cancer screening.
how introducing the option of HPV self-testing affects patient experience | Month 36
  Understand how introducing the option of non-invasive testing affects the patient experience for TGD patients undergoing hysterectomy. Recruited participants who are undergoing hysterectomy for gender-affirmation will be asked to complete surveys (N=30) and qualitative interviews (N=15) to evaluate how the option of self-testing or non-invasive testing affects the patient experience.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Wise, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneota, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No